CLINICAL TRIAL: NCT02676596
Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of K-312 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: K-312-1.02US
Record Dates: First submitted 2016-02-02; First posted 2016-02-08 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Other): Japanese and Non-Japanese subjects receiving K-312 50 mg QD
  Interventions: Drug: K-312 50 mg QD; Other: Placebo
- Cohort 2 (Other): Japanese and Non-Japanese subjects receiving K-312 100 mg QD
  Interventions: Drug: K-312 100 mg QD; Other: Placebo
- Cohort 3 (Other): Japanese and Non-Japanese subjects receiving K-312 200 mg QD
  Interventions: Drug: K-312 200 mg QD; Other: Placebo
- Cohort 4 (Other): Japanese and Non-Japanese subjects receiving K-312 400 mg QD
  Interventions: Drug: K-312 400 mg QD; Other: Placebo
- Cohort 5 (Other): Japanese and Non-Japanese subjects receiving K-312 25 mg QD
  Interventions: Drug: K-312 25 mg QD; Other: Placebo
- Cohort 6 (Other): Japanese and Non-Japanese subjects receiving K-312 10 mg QD
  Interventions: Drug: K-312 10 mg QD; Other: Placebo

INTERVENTIONS:
Drug: K-312 10 mg QD
  Arms: Cohort 6
Drug: K-312 25 mg QD
  Arms: Cohort 5
Drug: K-312 50 mg QD
  Arms: Cohort 1
Drug: K-312 100 mg QD
  Arms: Cohort 2
Drug: K-312 200 mg QD
  Arms: Cohort 3
Drug: K-312 400 mg QD
  Arms: Cohort 4
Other: Placebo

SUMMARY:
The purpose of this study is to investigate the safety tolerability, and PK profile of K-312 and its metabolites in healthy Japanese and non-Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male or a female of non-childbearing potential between the ages of 18 and 45 years, inclusive.
* Subject has a body mass index of 18.5 to 30 kg/m2, inclusive.
* Subject has hematology, coagulation, serum chemistry, and urinalysis test results within the reference ranges or showing no clinically relevant deviations, as judged by the Investigator.

Exclusion Criteria:

* Subject has the presence of an active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment.
* Subject has any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of K-312. Cholecystectomy is permitted if there are no postcholecystectomy gastrointestinal symptoms.
* Subject has clinically relevant abnormalities in clinical laboratory parameters.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
CETP activity | Days 1, 3, 6, 11, 16, 21, 27 and 30
Area under the plasma concentration | Days 1 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale, California, United States